CLINICAL TRIAL: NCT04814628
Title: Contribution of Transnasal Humidified Rapid-insufflation Ventilatory Exchange (THRIVE) to Optimize Maternal Pre-oxygenation and Anaesthetic Preparation Time for General Anaesthesia for Urgent Caesarean Section A Prospective Experimental Study on Healthy Volunteers.
Brief Title: Assessment of Transnasal Humidified Rapid-insufflation Ventilatory Exchange (THRIVE) for Maternal Pre-oxygenation
Acronym: PREOXCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL20_1116; 2021-A00047-34 (Other: ID-RCB)
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Cesarean Section Complications; Pregnancy Related; Anesthesia
Keywords: maternal preoxygenation; ventilatory exchange
MeSH Terms: interventions — Fees and Charges

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy volunteer subject (Experimental): A single healthy volunteer subject will participate in the study as a model of a pregnant woman in the third trimester of pregnancy, with a functional respiratory capacity reduced by 20% thanks to elastic restraints performed under the control of functional respiratory explorations.
  8 obstetric anesthesiologists will participate in the 4 scenarios;
  Interventions: Procedure: scenario 1 : pre-oxygenation with a face mask held by the anaesthetist; Procedure: scenario 2: one anaesthetist in charge, face mask held by the patient for pre-oxygenation; Procedure: scenario 3: one anaesthetist in charge, THRIVE used for pre-oxygenation; Procedure: scenario 4: one anaesthetist and one nurse anaesthetist in charge, the face mask is held by the anaesthetist or the nurse anaesthetist

INTERVENTIONS:
Procedure: scenario 1 : pre-oxygenation with a face mask held by the anaesthetist — the face mask is held by the anaesthetist (reference technique) to obtain effective pre-oxygenation for Oxygen Reserve Index (ORI) which has reached a plateau value for more than 10 seconds. All the usual supplies and medicines are available and in the same place as usual.
  The sequence is as follows:
  1. Patient lying on the operating table, start of the stopwatch
  2. Opening of the computerized anaesthesia file
  3. Monitoring (ECG, non-invasive blood pressure, SaO2) of the patient
  4. Preparation of the hypnotic (propofol or thiopental, as desired)
  5. Preparation of curare (succinylcholine or rocuronium, as desired)
  6. Pre-oxygenation of the patient with the face mask held by the participating anaesthetist
  7. Waiting for an ORI which has reached a plateau value for more than 10 seconds
  8. Conditions for general anaesthesia met for the participating anaesthetist
  9. "End of simulation", stopwatch stop
Procedure: scenario 2: one anaesthetist in charge, face mask held by the patient for pre-oxygenation — one anaesthetist is in charge of the simulated patient (volunteer), face mask held by the volunteer for pre-oxygenation for ORI which has reached a plateau value for more than 10 seconds All the usual supplies and medicines are available and in the same place as usual.
  The sequence is as follows:
  1. Patient entering the operating room, patient lying on the operating table, start of the stopwatch
  2. Opening of the computerized anaesthesia file
  3. Monitoring (ECG, non-invasive blood pressure, SaO2) of the patient
  4. Preparation of the hypnotic (propofol or thiopental, as desired)
  5. Preparation of curare (succinylcholine or rocuronium, as desired)
  6. Face mask held by the patient for pre-oxygenation
  7. Waiting for an ORI which has reached a plateau value for more than 10 seconds
  8. Conditions for general anaesthesia met for the participating anaesthetist
  9. "End of simulation", stopwatch stop
Procedure: scenario 3: one anaesthetist in charge, THRIVE used for pre-oxygenation — All the usual supplies and medicines are available and in the same place as usual.
  The sequence is as follows:
  1. Patient entering the operating room, patient lying on the operating table, start of the stopwatch
  2. Opening of the computerized anaesthesia file
  3. Monitoring (ECG, non-invasive blood pressure, SaO2) of the patient
  4. Preparation of the hypnotic (propofol or thiopental, as desired)
  5. Preparation of curare (succinylcholine or rocuronium, as desired)
  6. THRIVE for pre-oxygenation
  7. Waiting for an ORI which has reached a plateau value for more than 10 seconds
  8. Conditions for general anaesthesia met for the participating anaesthetist
  9. "End of simulation", stopwatch stop
Procedure: scenario 4: one anaesthetist and one nurse anaesthetist in charge, the face mask is held by the anaesthetist or the nurse anaesthetist — All the usual supplies and medicines are available and in the same place as usual.
  The sequence is as follows:
  1. Patient entering the operating room, patient lying on the operating table, start of the stopwatch
  2. Opening of the computerized anaesthesia file
  3. Monitoring (ECG, non-invasive blood pressure, SaO2) of the patient
  4. Preparation of the hypnotic (propofol or thiopental, as desired)
  5. Preparation of curare (succinylcholine or rocuronium, as desired)
  6. Pre-oxygenation of the patient with the face mask held by the participating anaesthetist or nurse anaesthetist
  7. Waiting for an ORI which has reached a plateau value for more than 10 seconds
  8. Conditions for general anaesthesia met for the participating anaesthetist
  9. "End of simulation", stopwatch stop

SUMMARY:
The main objective of this study is to determine if the use of transnasal humidified rapid-insufflation ventilatory exchange (THRIVE) can reduce by 90 seconds the time between the entry into the operating room of the volunteer and the moment when the anaesthetic drugs are ready and when the Oxygen Reserve Index has reached a plateau value for more than 10 seconds, a moment which would therefore allow the induction of general anaesthesia, compared to the pre-oxygenation with the face mask applied by the anaesthetist alone in charge of anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* major
* female
* affiliated to a social security scheme or beneficiary of such a scheme
* having voluntarily and informedly agreed to participate in the study.
* non-smoker
* free from pulmonary, cardiac and neurological pathologies
* have a normal functional respiratory test at baseline.

Exclusion Criteria:

* refusal to participate in the study
* non-French speaking volunteer
* obesity defined by a body mass index greater than 30 kilogram/meter² (kg/m²)
* current pregnancy
* Volunteer in period of exclusion from further research
* Person under guardianship, curatorship or any other administrative or judicial measure of deprivation of rights and liberty

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
time between when the volunteer enters the operating room and when the conditions for general anesthesia are met during pre-oxygenation | through study completion, an average of 1 year
  Difference between the time when volunteer enters the operating room and the time when the conditions for general anaesthesia are met during pre-oxygenation with the face mask applied by one anaesthesist in charge of the volunteer (simulated patient) compared to the use of preoxygenation with THRIVE by one anaesthesist in charge of the volunteer

SECONDARY OUTCOMES:
time between volunteer enters the operating room and when the conditions for general anaesthesia are met during pre-oxygenation | through study completion, an average of 1 year
  Difference between the time when volunteer enters the operating room and the time when the conditions for general anaesthesia are met during pre-oxygenation with the face mask applied by one anaesthetist in charge of the volunteer (simulated patient), during pre-oxygenation with the face mask applied by the volunteer (one anaesthetist in charge of the simulated patient), during preoxygenation with THRIVE (one anaesthetist in charge of the simulated patient), during preoxygenation with the facemask applied by the anaesthetist or the nurse anaesthetist both in charge of the simulated patient
number of medication errors during the preparation | through study completion, an average of 1 year
  Medication errors occurring during treatment in the 4 scenarios will be counted (medication preparation errors, no medication is administered to the volunteer)
number of deviations from appropriate anaesthetic practices observed during preparation | through study completion, an average of 1 year
  The number of deviations from the appropriate anesthetic practices observed during the preparation will be counted in the 4 scenarios

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Femme Mère Enfant, Bron, France